CLINICAL TRIAL: NCT04562818
Title: Results From a Mexican Long-term Multicentric Study on Acute Promyelocytic Leukemia.
Brief Title: Results From a Mexican Acute Promyelocytic Leukemia.
Acronym: Mexico APL
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Nidia Paulina Zapata-Canto, Assistant Professor of Hematology Department (Acute Myeloid Leukemia), Instituto Nacional de Cancerologia de Mexico
Other Study IDs: INCancerologiaMexico
Record Dates: First submitted 2020-06-08; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Promyelocytic Leukemia, Acute
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Diagnosis; Karyotype; Leukocyte Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Daunorrubicin: Patient treated with daunorrubicin
  Interventions: Diagnostic Test: Diagnosis; Diagnostic Test: Molecular and Karyotype; Diagnostic Test: Leucocytes
- Idarrubicin: Patient treated with idarrubicin
  Interventions: Diagnostic Test: Diagnosis; Diagnostic Test: Molecular and Karyotype; Diagnostic Test: Leucocytes

INTERVENTIONS:
Diagnostic Test: Diagnosis — Determine the number of center that are able to process PCR or FISH/Karyotype for PML/RAR or t(15;17)
Diagnostic Test: Molecular and Karyotype — To realize the need of having more center we the technology to perform all of these tests
  Other Names: FISH; Karyotype; PCR
Diagnostic Test: Leucocytes
  Other Names: Risk status

SUMMARY:
Retrospective, observational study, comparing treatments of acute promyelocytic leukemia in different centers in México.

There is no sufficient information about acute promyelocytic leukemia in America Latina, particularly in Mexico.

For these reason the investigators started a study adding all promyelocityc patients from the main Hospital in Mexico in order to put together a group of patient and analyze the response, overall survival and what are the characteristics of the population.

The investigators included 5 Hospital in Mexico City and states as Monterrey, Guadalajara, San Luis Potosi, Puebla, Veracruz, Yucatán, Oaxaca, Guanajuato, Estado de México.

Even do, the investigators didn´t have arsenic trioxide they are treating patients with standard chemotherapy. These paper will help to show the authorities that the cost of treating patient with standard chemotherapy is much more higher than ATO-ATRA. The investigators are now doing a cost benefit analysis so the investigators, can soon have ATO treatment as standard of care in Mexico for the treatment of acute promyelocytic leukemia.

DETAILED DESCRIPTION:
A multicentric, retrospective, descriptive, longitudinal study was carried out. Between January 2007 and January 2017, patients of both sexes and different ages, who were candidates for receiving intensive chemotherapy along with tretinoin were included in the study. The diagnosis for Acute Promyelocytic Leukemia was determined based on the following criteria: abnormal promyelocytes in the bone marrow and verification of the t(15;17) translocation by karyotype or using RT-PCR to determine the genetic lesion and define the type of PML/RARA isoform.

In Mexico the investigators still treating patients with anthracycline and cytarabine + transretinoic acid. These information will help the authorities to realize the importance of having arsenic trioxide as part of the treatment of these disease, knowing the amount of patient that the investigators have in Mexico, knowing that in the hispanic race the incidence is greater.

ELIGIBILITY:
Inclusion Criteria:

* Actute Promyelocytic leukemia PML/RAR alfa + Diabetes mellitus Hypertension Asthma Chronic renal disease

Exclusion Criteria:

* Non Acute Promyelocytic leukemia Younger than 15 years old

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient older 15 years old with acute promyelocytic Leukemia treated at a Mecican Center
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival in Mexico in patients with acute promyelocytic leukemia | January 2007- January 2017
  Overall survival in different institutions in Mexico, in patient with diagnostic with acute promyelocytic leukemia

SECONDARY OUTCOMES:
Difference in survival with different anthracycline (Daunorrubicin vs idarrubicin) | January 2007-January 2017
  Event free survival and overall survival with different anthracyclin
Complications with different anthracycline | January 2007-January 2017
  Complications

CONTACTS AND LOCATIONS:
Locations (1):
- Nidia Zapata, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Plan is to published the information in Mexico, so we can start planing with the Mexican government the cost of treating a patient with Chemotherapy vs ATO/ATRA

REFERENCES:
- [Result] Sanz MA, Fenaux P, Tallman MS, Estey EH, Lowenberg B, Naoe T, Lengfelder E, Dohner H, Burnett AK, Chen SJ, Mathews V, Iland H, Rego E, Kantarjian H, Ades L, Avvisati G, Montesinos P, Platzbecker U, Ravandi F, Russell NH, Lo-Coco F. Management of acute promyelocytic leukemia: updated recommendations from an expert panel of the European LeukemiaNet. Blood. 2019 Apr 11;133(15):1630-1643. doi: 10.1182/blood-2019-01-894980. Epub 2019 Feb 25. PMID 30803991
- [Result] Cicconi L, Fenaux P, Kantarjian H, Tallman M, Sanz MA, Lo-Coco F. Molecular remission as a therapeutic objective in acute promyelocytic leukemia. Leukemia. 2018 Aug;32(8):1671-1678. doi: 10.1038/s41375-018-0219-5. Epub 2018 Jul 19. PMID 30026570
- [Result] Ryan MM. Acute Promyelocytic Leukemia: A Summary. J Adv Pract Oncol. 2018 Mar;9(2):178-187. Epub 2018 Mar 1. PMID 30588352
- [Result] Warrell RP Jr, de The H, Wang ZY, Degos L. Acute promyelocytic leukemia. N Engl J Med. 1993 Jul 15;329(3):177-89. doi: 10.1056/NEJM199307153290307. PMID 8515790
- [Result] Barbui T, Finazzi G, Falanga A. The impact of all-trans-retinoic acid on the coagulopathy of acute promyelocytic leukemia. Blood. 1998 May 1;91(9):3093-102. No abstract available. PMID 9558362
- [Result] Tallman MS, Kwaan HC. Reassessing the hemostatic disorder associated with acute promyelocytic leukemia. Blood. 1992 Feb 1;79(3):543-53. No abstract available. PMID 1732003
- [Result] Fenaux P, Le Deley MC, Castaigne S, Archimbaud E, Chomienne C, Link H, Guerci A, Duarte M, Daniel MT, Bowen D, et al. Effect of all transretinoic acid in newly diagnosed acute promyelocytic leukemia. Results of a multicenter randomized trial. European APL 91 Group. Blood. 1993 Dec 1;82(11):3241-9. PMID 8241496
- [Result] Krutova TV, Linchina LP, Korman DB, Isaev NM, Shkrob OS. [Autoradiographic study of the gastric mucosa in cancer]. Vopr Onkol. 1976;22(10):8-13. Russian. PMID 189506
- [Result] Licht JD, Chomienne C, Goy A, Chen A, Scott AA, Head DR, Michaux JL, Wu Y, DeBlasio A, Miller WH Jr, et al. Clinical and molecular characterization of a rare syndrome of acute promyelocytic leukemia associated with translocation (11;17). Blood. 1995 Feb 15;85(4):1083-94. PMID 7849296
- [Result] Arber DA, Orazi A, Hasserjian R, et al. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016;127(20):2391-2405. Blood. 2016 Jul 21;128(3):462-463. doi: 10.1182/blood-2016-06-721662. No abstract available. PMID 31659364
- [Result] Avvisati G, Lo-Coco F, Paoloni FP, Petti MC, Diverio D, Vignetti M, Latagliata R, Specchia G, Baccarani M, Di Bona E, Fioritoni G, Marmont F, Rambaldi A, Di Raimondo F, Kropp MG, Pizzolo G, Pogliani EM, Rossi G, Cantore N, Nobile F, Gabbas A, Ferrara F, Fazi P, Amadori S, Mandelli F; GIMEMA, AIEOP, and EORTC Cooperative Groups. AIDA 0493 protocol for newly diagnosed acute promyelocytic leukemia: very long-term results and role of maintenance. Blood. 2011 May 5;117(18):4716-25. doi: 10.1182/blood-2010-08-302950. Epub 2011 Mar 8. PMID 21385856
- [Result] Powell BL, Moser B, Stock W, Gallagher RE, Willman CL, Stone RM, Rowe JM, Coutre S, Feusner JH, Gregory J, Couban S, Appelbaum FR, Tallman MS, Larson RA. Arsenic trioxide improves event-free and overall survival for adults with acute promyelocytic leukemia: North American Leukemia Intergroup Study C9710. Blood. 2010 Nov 11;116(19):3751-7. doi: 10.1182/blood-2010-02-269621. Epub 2010 Aug 12. PMID 20705755
- [Result] Platzbecker U, Avvisati G, Cicconi L, Thiede C, Paoloni F, Vignetti M, Ferrara F, Divona M, Albano F, Efficace F, Fazi P, Sborgia M, Di Bona E, Breccia M, Borlenghi E, Cairoli R, Rambaldi A, Melillo L, La Nasa G, Fiedler W, Brossart P, Hertenstein B, Salih HR, Wattad M, Lubbert M, Brandts CH, Hanel M, Rollig C, Schmitz N, Link H, Frairia C, Pogliani EM, Fozza C, D'Arco AM, Di Renzo N, Cortelezzi A, Fabbiano F, Dohner K, Ganser A, Dohner H, Amadori S, Mandelli F, Ehninger G, Schlenk RF, Lo-Coco F. Improved Outcomes With Retinoic Acid and Arsenic Trioxide Compared With Retinoic Acid and Chemotherapy in Non-High-Risk Acute Promyelocytic Leukemia: Final Results of the Randomized Italian-German APL0406 Trial. J Clin Oncol. 2017 Feb 20;35(6):605-612. doi: 10.1200/JCO.2016.67.1982. Epub 2016 Oct 31. PMID 27400939
- [Result] Hiorns LR, Swansbury GJ, Mehta J, Min T, Dainton MG, Treleaven J, Powles RL, Catovsky D. Additional chromosome abnormalities confer worse prognosis in acute promyelocytic leukaemia. Br J Haematol. 1997 Feb;96(2):314-21. doi: 10.1046/j.1365-2141.1997.d01-2037.x. PMID 9029019
- [Result] Iland HJ, Bradstock K, Supple SG, Catalano A, Collins M, Hertzberg M, Browett P, Grigg A, Firkin F, Hugman A, Reynolds J, Di Iulio J, Tiley C, Taylor K, Filshie R, Seldon M, Taper J, Szer J, Moore J, Bashford J, Seymour JF; Australasian Leukaemia and Lymphoma Group. All-trans-retinoic acid, idarubicin, and IV arsenic trioxide as initial therapy in acute promyelocytic leukemia (APML4). Blood. 2012 Aug 23;120(8):1570-80; quiz 1752. doi: 10.1182/blood-2012-02-410746. Epub 2012 Jun 19. PMID 22715121
- [Result] Grimwade D, Walker H, Oliver F, Wheatley K, Harrison C, Harrison G, Rees J, Hann I, Stevens R, Burnett A, Goldstone A. The importance of diagnostic cytogenetics on outcome in AML: analysis of 1,612 patients entered into the MRC AML 10 trial. The Medical Research Council Adult and Children's Leukaemia Working Parties. Blood. 1998 Oct 1;92(7):2322-33. PMID 9746770
- [Result] De Botton S, Chevret S, Sanz M, Dombret H, Thomas X, Guerci A, Fey M, Rayon C, Huguet F, Sotto JJ, Gardin C, Cony Makhoul P, Travade P, Solary E, Fegueux N, Bordessoule D, San Miguel J, Link H, Desablens B, Stamatoullas A, Deconinck E, Geiser K, Hess U, Maloisel F, Castaigne S, Preudhomme C, Chomienne C, Degos L, Fenaux P; European APL Group. Additional chromosomal abnormalities in patients with acute promyelocytic leukaemia (APL) do not confer poor prognosis: results of APL 93 trial. Br J Haematol. 2000 Dec;111(3):801-6. doi: 10.1046/j.1365-2141.2000.02442.x. PMID 11122141